CLINICAL TRIAL: NCT01365663
Title: A First-in-Human (FIH), Randomized, Dose-Escalation, Double-Blind, Placebo-Controlled Study to Assess Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of SPC4955 Administered to Healthy Subjects
Brief Title: Multiple Ascending Dose Study of SPC4955 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santaris Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPC4955-901; EudraCT 2010-024363-40
Record Dates: First submitted 2011-05-18; First posted 2011-06-03 (Estimated); Last update posted 2012-01-31 (Estimated); Status verified 2012-01

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; LDL; HDL; apoB; hyperlipidemia; LNA-oligonucleotide
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cohort 1 (Experimental): 0.25 mg/kg in Healthy Subjects
  Interventions: Drug: SPC4955
- Cohort 2 (Experimental): 0.5 mg/kg in Healthy Subjects
  Interventions: Drug: SPC4955
- Cohort 3 (Experimental): 1.0 mg/kg in Healthy Subjects
  Interventions: Drug: SPC4955
- Cohort 4 (Experimental): 1.5 mg/kg in Healthy Subjects
  Interventions: Drug: SPC4955
- Cohort 5 (Experimental): 2.0 mg/kg in Healthy Subjects
  Interventions: Drug: SPC4955
- Saline 0.9% (Placebo Comparator)
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: SPC4955 — 3 Weekly SC injections
  Arms: Cohort 1
Drug: SPC4955 — 3 Weekly SC injections
  Arms: Cohort 2
Drug: SPC4955 — 3 Weekly SC injections
  Arms: Cohort 3
Drug: SPC4955 — 3 Weekly SC injections
  Arms: Cohort 4
Drug: SPC4955 — 3 Weekly SC injections
  Arms: Cohort 5
Drug: Saline 0.9% — 3 Weekly SC injections
  Arms: Saline 0.9%

SUMMARY:
The purpose of this study is to study safety and tolerability of SPC4955 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, age 18-65 years, inclusive.
2. BMI 18-33 kg/m2
3. Screening hematology, clinical chemistries, coagulation and urinalysis consistent with overall good health and the following criteria are met:

   * LDL-C ≥3.24 mmol/L (≥125 mg/dL)
   * Triglycerides (fasted) <2.7mmol/L (<239 mg/dL)
   * ALT within normal limits

Exclusion Criteria:

1. Any uncontrolled or active major systemic disease including, but not limited to: cardiovascular, pulmonary, gastrointestinal, metabolic, urogenital, neurological, immunological, psychiatric, or neoplastic disorder with metastatic potential.
2. History or presence of malignancy within the past year. Subjects who have been successfully treated (for 3 months or longer) with no recurrence of basal cell carcinoma of the skin or carcinoma in-situ of the cervix may be enrolled
3. Active acute or chronic infection, including, but not limited to: upper airway infection, urinary tract infection, and skin infection
4. Use of prescription medication within 14 days prior to the planned first drug administration and throughout the study.
5. Use of non-prescription or over-the-counter medications is prohibited within 7 days prior to the planned first drug administration and throughout the study. This includes all vitamins, herbal supplements, or remedies.
6. Positive results on the following Screening laboratory tests: urine pregnancy test (women only), alcohol breath test, urine drugs of abuse, hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV) antibody.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-05; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects experiencing adverse events | up to 78 days

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of SPC4955 | Up to 78 Days
total Cholesterol | up to 78 days
Area under the plasma concentration versus time curve (AUC) of SPC4955 | Up to 78 days
LDL | up to 78 days
HDL | up to 78 days

CONTACTS AND LOCATIONS:
Overall Officials: Werner Feuerer, Dr. med., Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany